CLINICAL TRIAL: NCT02296320
Title: A Phase 2 Randomised, Double-blind, Placebo-controlled, Single-dose, Dose-ranging Study of the Efficacy and Safety of MEDI4893, a Human Monoclonal Antibody Against Staphylococcus Aureus Alpha Toxin in Mechanically Ventilated Adult Subjects.
Brief Title: Study of the Efficacy and Safety of MEDI4893
Acronym: SAATELLITE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Innovative Medicines Initiative (Other); Antibacterial Resistance Leadership Group (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CD-ID-MEDI4893-1139
Record Dates: First submitted 2014-10-30; First posted 2014-11-20 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Staphylococcus Aureus Pneumonia
MeSH Terms: conditions — Pneumonia, Staphylococcal | interventions — suvratoxumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MEDI4893 5000 mg (Active Comparator): Participants will receive a single intravenous (IV) dose of MEDI4893 5000 milligrams (mg) on Day 1 of the study.
  Interventions: Drug: MEDI4893
- Placebo (Placebo Comparator): Participants will receive a single IV dose of placebo matched to MEDI4893 on Day 1 of the study.
  Interventions: Other: Placebo
- MEDI4893 2000 mg (Active Comparator): Participants will receive a single IV dose of MEDI4893 2000 mg on Day 1 of the study.
  Interventions: Drug: MEDI4893

INTERVENTIONS:
Drug: MEDI4893 — Participants will receive a single IV dose of MEDI4893 2000 or 5000 mg on Day 1 of the study.
  Arms: MEDI4893 2000 mg; MEDI4893 5000 mg
Other: Placebo — Participants will receive a single IV dose of placebo matched to MEDI4893 on Day 1 of the study.
  Arms: Placebo

SUMMARY:
Clinical trial looking at safety and efficacy of MEDI4893 in prevention of pneumonia caused by Staphylococcus aureus in high-risk patients

ELIGIBILITY:
Inclusion Criteria:

* Colonized with Staphylococcus aureus, expected to require prolonged intubation and mechanical ventilation, without any evidence of active pneumonia.

Exclusion Criteria:

* Staphylococcal disease at randomisation; lung injury score consistent with pneumonia; current lung disease; chronic tracheostomy patients; currently receiving systemic anti-staphylococcal antibiotics; moribund patients.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2014-10-10 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (45):
- United States (2):
  - Research Site, Atlanta, Georgia
  - Research Site, Detroit, Michigan
- Belgium (5):
  - Research Site, Arlon
  - Research Site, Brussels
  - Research Site, La Louvière
  - Research Site, Lodelinsart
  - Research Site, Yvoir
- Czechia (5):
  - Research Site, Brno
  - Research Site, Děčín
  - Research Site, Kyjov
  - Research Site, Prague
  - Research Site, Teplice
- France (14):
  - Research Site, Angers
  - Research Site, Clermont-Ferrand
  - Research Site, Garches
  - Research Site, Grenoble
  - Research Site, Le Chesnay
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Nantes
  - Research Site, Orléans
  - Research Site, Pierre-Bénite
  - Research Site, Poitiers
  - Research Site, Rennes
  - Research Site, Tours
- Germany (4):
  - Research Site, Berlin
  - Research Site, Erfurt
  - Research Site, Heidelberg
  - Research Site, Jena
- Greece (4):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Ioannina
  - Research Site, Larissa
- Hungary (2):
  - Research Site, Kistarcsa
  - Research Site, Vác
- Research Site, Ponte de Lima, Portugal
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Getafe
  - Research Site, Madrid
  - Research Site, Oviedo
  - Research Site, Terrassa
  - Research Site, Valencia
- Switzerland (2):
  - Research Site, Geneva
  - Research Site, Lausanne

REFERENCES:
- [Derived] Francois B, Jafri HS, Chastre J, Sanchez-Garcia M, Eggimann P, Dequin PF, Huberlant V, Vina Soria L, Boulain T, Bretonniere C, Pugin J, Trenado J, Hernandez Padilla AC, Ali O, Shoemaker K, Ren P, Coenjaerts FE, Ruzin A, Barraud O, Timbermont L, Lammens C, Pierre V, Wu Y, Vignaud J, Colbert S, Bellamy T, Esser MT, Dubovsky F, Bonten MJ, Goossens H, Laterre PF; COMBACTE Consortium and the SAATELLITE Study Group. Efficacy and safety of suvratoxumab for prevention of Staphylococcus aureus ventilator-associated pneumonia (SAATELLITE): a multicentre, randomised, double-blind, placebo-controlled, parallel-group, phase 2 pilot trial. Lancet Infect Dis. 2021 Sep;21(9):1313-1323. doi: 10.1016/S1473-3099(20)30995-6. Epub 2021 Apr 21. PMID 33894131
- [Derived] Yu XQ, Robbie GJ, Wu Y, Esser MT, Jensen K, Schwartz HI, Bellamy T, Hernandez-Illas M, Jafri HS. Safety, Tolerability, and Pharmacokinetics of MEDI4893, an Investigational, Extended-Half-Life, Anti-Staphylococcus aureus Alpha-Toxin Human Monoclonal Antibody, in Healthy Adults. Antimicrob Agents Chemother. 2016 Dec 27;61(1):e01020-16. doi: 10.1128/AAC.01020-16. Print 2017 Jan. PMID 27795368
- See also: CD-ID-MEDI4893-1139 Protocol amendment 5_redacted_FINAL_APPROVED — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CD-ID-MEDI4893-1139&attachmentIdentifier=516e4676-ac10-48ef-8f1b-f2c3bacfc92f&fileName=CD-ID-MEDI4893-1139_Protocol_amendment_5_redacted_FINAL_APPROVED.pdf&versionIdentifier=
- See also: CD-ID-MEDI4893-1139 Statistical Analysis Plan_Final v4.0_Redacted_FINAL_APPROVED — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CD-ID-MEDI4893-1139&attachmentIdentifier=3b2d9a7a-eaa9-4651-be9d-7271be664bb1&fileName=CD-ID-MEDI4893-1139_Statistical_Analysis_Plan_Final_v4.0_Redacted_FINAL_APPROVED.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 10Oct2014 and 02Oct2018.
Pre-assignment Details: A total of 767 participants consented to participate in the study, of which 554 were screen failures. A total of 213 participants were randomized in the study.
Groups:
- Placebo: Participants received a single IV dose of placebo matched to MEDI4893 on Day 1 of the study.
- MEDI4893 2000 mg: Participants received a single IV dose of MEDI4893 2000 milligrams (mg) on Day 1 of the study.
- MEDI4893 5000 mg: Participants received a single IV dose of MEDI4893 5000 mg on Day 1 of the study.
Period: Overall Study
Arm/Group | Placebo | MEDI4893 2000 mg | MEDI4893 5000 mg
Started | 102 | 15 | 96
Treated | 100 | 15 | 96
Completed | 67 | 10 | 59
Not Completed | 35 | 5 | 37
Not completed — Withdrawal by Subject | 4 | 0 | 2
Not completed — Death | 24 | 3 | 27
Not completed — Lost to Follow-up | 5 | 2 | 7
Not completed — Not treated | 2 | 0 | 0
Not completed — Not - specified | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-treat (mITT) population included all participants, who received any dose of study drug and analyzed according to their randomized treatment group.
Groups:
- MEDI4893 2000 mg: Participants received a single IV dose of MEDI4893 2000 mg on Day 1 of the study.
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI4893 2000 mg | MEDI4893 5000 mg | Total
Number analyzed (Participants) | 100 | 15 | 96 | 211
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (16.6) | 52.5 (14.6) | 57.7 (15.7) | 56.4 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 5 | 37 | 87
  Male | 55 | 10 | 59 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4 | 8
  Not Hispanic or Latino | 96 | 15 | 92 | 203
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 2 | 6
  White | 97 | 13 | 94 | 204
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Endpoint Adjudication Committee-Determined (EAC) Staphylococcus Aureus (S Aureus) Pneumonia
Description: The EAC S aureus pneumonia was based on clinical, radiographic, and microbiologic criteria. Clinical criteria: 1 major criteria (PaO2/FiO2 ratio < 240 mmHg maintained for at least 4 hours or decrease in PaO2/FiO2 by >= 50 mmHg maintained for at least 4 hrs or a need to initiate non-invasive mechanical ventilation or re-initiate invasive mechanical ventilation because of respiratory failure or worsening of respiratory status); and at least 2 of minor criteria (systemic signs of infection, production of purulent sputum/endotracheal secretions, new onset of cough, physical examination findings consistent with pneumonia/pulmonary consolidation, dyspnea, and/or tachypnea). Radiographic criteria: new or worsening infiltrate consistent with pneumonia on chest X-ray obtained within 24 hrs of event. Microbiologic criteria: at least 1 culture positive for S aureus (respiratory specimen, or blood, or pleural fluid aspirate or lung tissue culture during episode of pneumonia).
Time Frame: Day 1 through Day 31
Population: An mITT population included all participants, who received any dose of study drug and analyzed according to their randomized treatment group.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | MEDI4893 2000 mg | MEDI4893 5000 mg
Number analyzed (Participants) | 100 | 15 | 96
Percentage of Participants | 26.0 | 20.0 | 17.7
Statistical Analysis 1: Comparison: Placebo vs MEDI4893 5000 mg; The key efficacy analyses were based on 5000 mg MEDI4893 and placebo. Participants who received 2000 mg MEDI4893 were summarized descriptively; Test type: Superiority; p = 0.166, Poisson regression with robust variance; Relative risk reduction = 31.9, 90% CI 2-sided [-7.5 to 56.8]

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Through 31 Days
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through Day 31
Population: As-treated population included all participants, who received any dose of study drug and analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI4893 2000 mg | MEDI4893 5000 mg
Number analyzed (Participants) | 100 | 15 | 96
Participants | 90 | 15 | 87

3. Primary Outcome: Number of Participants With TEAEs Through 91 Days
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through Day 91
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI4893 2000 mg | MEDI4893 5000 mg
Number analyzed (Participants) | 100 | 15 | 96
Participants | 92 | 15 | 89

4. Primary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (TESAEs)
Description: A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through Day 191
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI4893 2000 mg | MEDI4893 5000 mg
Number analyzed (Participants) | 100 | 15 | 96
Participants | 40 | 7 | 50

5. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: An AESI is one of scientific and medical interest specific to understanding of the study drug and may have required close monitoring and rapid communication by the investigator to the sponsor. An AESI may have been serious or non-serious.
Time Frame: Day 1 through Day 191
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI4893 2000 mg | MEDI4893 5000 mg
Number analyzed (Participants) | 100 | 15 | 96
Participants | 0 | 4 | 3

6. Primary Outcome: Number of Participants With New Onset Chronic Diseases (NOCDs)
Description: An NOCD defined as a newly diagnosed medical condition that is of a chronic, ongoing nature. It is observed after receiving the study drug and is assessed by the investigator as medically significant.
Time Frame: Day 1 through Day 191
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI4893 2000 mg | MEDI4893 5000 mg
Number analyzed (Participants) | 100 | 15 | 96
Participants | 2 | 0 | 3

7. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of MEDI4893
Description: Maximum observed serum concentration (Cmax) of MEDI4893 is reported.
Time Frame: Day 1 (Pre-dose, end of the infusion, 8 and 24 hours post dose), and on Days 4, 8, 15, 22, 31, 61, and 91
Population: An Intent-to-treat (ITT) population included all randomized participants and were analyzed according to their randomized treatment group. Participants who had quantifiable pharmacokinetic (PK) samples were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | MEDI4893 2000 mg | MEDI4893 5000 mg
Number analyzed (Participants) | 14 | 94
μg/mL | 471.9 (123.0) | 1143.7 (375.6)

8. Secondary Outcome: Area Under the Serum Concentration Time Curve From Time Zero to Last Measurable Concentration (AUC [0-Last]) of MEDI4893
Description: Area under the serum concentration time curve from time zero to last measurable concentration (AUC[0 - Last]) of MEDI4893 is reported.
Time Frame: Day 1 (Pre-dose, end of the infusion, 8 and 24 hours post dose), and on Days 4, 8, 15, 22, 31, 61, and 91
Population: An ITT population included all randomized participants and were analyzed according to their randomized treatment group. Participants who had quantifiable PK samples were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | MEDI4893 2000 mg | MEDI4893 5000 mg
Number analyzed (Participants) | 14 | 94
day*μg/mL | 9045.5 (5383.1) | 20127.5 (12852.2)

9. Secondary Outcome: Observed Serum Concentration of MEDI4893 Through 30 Days Post Dose (C30)
Description: Observed serum concentration of MEDI4893 through 30 days post dose (C30) is reported. Serum concentration of MEDI4893 through 30 days post dose accounted the overall concentration of MEDI4893 measured on specified time points (Days 1, 4, 8, 15, 22, and 30).
Time Frame: Day 1 (Pre-dose, end of the infusion, 8 and 24 hours post dose), and on Days 4, 8, 15, 22, and 30
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | MEDI4893 2000 mg | MEDI4893 5000 mg
Number analyzed (Participants) | 13 | 68
μg/mL | 122.0 (65.0) | 295.9 (130.6)

10. Secondary Outcome: Observed Serum Concentration of MEDI4893 Through 90 Days Post Dose (C90)
Description: Observed serum concentration of MEDI4893 through 90 days post dose (C90) is reported. Serum concentration of MEDI4893 through 90 days post dose accounted the overall concentration of MEDI4893 measured on specified time points (Days 1, 4, 8, 15, 22, 31, 61, and 91).
Time Frame: Day 1 (Pre-dose, end of the infusion, 8 and 24 hours post dose), and on Days 4, 8, 15, 22, 31, 61, and 90
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | MEDI4893 2000 mg | MEDI4893 5000 mg
Number analyzed (Participants) | 11 | 54
μg/mL | 71.5 (35.5) | 192.0 (84.0)

11. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) Titer to MEDI4893
Description: Participants with ADA-positive at any of Day 31, Day 61, or Day 91 post-baseline assessments were always counted as "positive" at post-baseline.
Time Frame: Pre-dose on Day 1 (Baseline); and on Days 31, 61, and 91
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI4893 2000 mg | MEDI4893 5000 mg
Number analyzed (Participants) | 100 | 15 | 96
Participants
  Positive at baseline | 3 | 0 | 2
  Positive post-baseline | 5 | 0 | 0
  Positive at baseline and post-baseline | 2 | 0 | 0
  Not detected at baseline; positive post-baseline | 3 | 0 | 0
  Positive at baseline; not detected post-baseline | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: SAEs: Day 1 through Day 191 AEs: Day 1 through Day 91
Arm/Group | Placebo | MEDI4893 2000 mg | MEDI4893 5000 mg
All-Cause Mortality (participants affected / at risk) | 24/100 | 3/15 | 27/96
Serious Adverse Events (participants affected / at risk) | 40/100 | 7/15 | 50/96
Other Adverse Events (participants affected / at risk) | 90/100 | 15/15 | 85/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=100) | MEDI4893 2000 mg (N=15) | MEDI4893 5000 mg (N=96)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Brain death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Acinetobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Creutzfeldt-jakob disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia serratia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Serratia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Serratia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Weaning failure (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1)
Coma scale abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Brain hypoxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Brain stem stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Coma (Nervous system disorders) | 1 (1) | 1 (2) | 5 (5)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Hypercapnic coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Multiple system atrophy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Nervous system disorder (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neurological decompensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (2)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 5 (5)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=100) | MEDI4893 2000 mg (N=15) | MEDI4893 5000 mg (N=96)
Anaemia (Blood and lymphatic system disorders) | 12 (24) | 2 (2) | 11 (11)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Normochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 6 (6)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1) | 2 (2)
Atrial flutter (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 3 (3) | 0 (0) | 3 (3)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular dystrophy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Right-to-left cardiac shunt (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 15 (16) | 1 (1) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 8 (11) | 3 (4) | 8 (13)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (4)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 0 (0) | 1 (1)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (5)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (6) | 0 (0) | 0 (0)
Catheter site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1)
Generalised oedema (General disorders) | 3 (3) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 3 (4) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Implant site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Medical device site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 15 (26) | 2 (5) | 8 (9)
Vascular complication associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1)
Biliary cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 4 (4) | 4 (4) | 7 (7)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 2 (3) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 5 (5) | 4 (4) | 6 (6)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Abscess bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Acinetobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Bacterial disease carrier (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bacteroides bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 5 (6) | 0 (0) | 2 (2)
Bronchitis pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Citrobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Citrobacter sepsis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 2 (4) | 0 (0) | 2 (2)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterobacter infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Enterobacter pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 14 (18) | 4 (4) | 18 (23)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Haemophilus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Klebsiella infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Moraxella infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Morganella infection (Infections and infestations) | 3 (5) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 17 (17) | 1 (1) | 7 (7)
Pneumonia escherichia (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia moraxella (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Pneumonia serratia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 13 (13) | 2 (2) | 13 (13)
Postoperative wound infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Proteus infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pseudomonas bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Puncture site abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Serratia bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Serratia infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 6 (7) | 1 (1) | 3 (3)
Staphylococcal infection (Infections and infestations) | 4 (5) | 0 (0) | 4 (4)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Systemic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (4)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Urinary tract infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 3 (3) | 1 (1) | 4 (4)
Urinary tract infection staphylococcal (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection bacterial (Infections and infestations) | 2 (2) | 0 (0) | 3 (3)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Eschar (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Mechanical ventilation complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Traumatic shock (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Unintentional medical device removal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Weaning failure (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (3) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Mononucleosis heterophile test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pancreatic enzymes increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cerebral salt-wasting syndrome (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 2 (2)
Hyperlactacidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (9) | 1 (2) | 11 (13)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 1 (1) | 4 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (4)
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin k deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Amyotrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (3)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic hyperosmolar coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 2 (3)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglossal nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Multiple system atrophy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle tone disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myoclonic epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Neurological decompensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Quadriplegia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Subdural hygroma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vasculitis cerebral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vocal cord paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 3 (4) | 0 (0) | 6 (6)
Anxiety (Psychiatric disorders) | 5 (5) | 1 (1) | 8 (8)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1) | 5 (7)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 1 (1) | 4 (4)
Flat affect (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1) | 5 (5)
Organic brain syndrome (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Male genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1) | 7 (7)
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 1 (1) | 0 (0)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Laryngeal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngeal granuloma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 1 (1)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0) | 6 (6)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haemodynamic instability (Vascular disorders) | 1 (3) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 8 (8) | 1 (1) | 7 (7)
Hypotension (Vascular disorders) | 2 (3) | 1 (2) | 7 (10)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Medimmune has 60 days to review results communications prior to public release and may delete information that compromises on-going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT02296320/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT02296320/SAP_001.pdf